CLINICAL TRIAL: NCT06616792
Title: Dexamethasone Phonophoresis Versus Laser Acupuncture on Chronic Rhinosinusitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Abd Elaziem Abd Elaziz, Walaa Abd Elaziem Abd Elaziz, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005254
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-06

CONDITIONS: Chronic Rhinosinusitis (CRS)
Keywords: Dexamethasone Phonophoresis, Laser Acupuncture, Chronic Rhinosinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group (A) (Experimental): Each participant in this group will receive dexamethasone phonophoresis, US with the use of 0.4% Dexamethasone sodium phosphate gel for phonophoresis. over maxillary and frontal sinuses for 3 sessions per week for one month, in addition to the traditional medication.
  Interventions: Combination Product: Dexamethasone phonophoresis; Other: Traditional medication
- Group (B) (Experimental): Each participant in this group will receive low level laser placed in contact with the skin perpendicular over the body acupoints (LI 4) - (LI 20) - (EX- HN5) - (GV 20) - (GV 24) - (ST3) - (ST 7) in both sides and on (EX-HN3) acupoint, with a duration of 90 sec for each point three times per week for a month., in addition to the traditional medication.
  Interventions: Device: Laser Acupuncture; Other: Traditional medication
- Group (C) (Active Comparator): Each participant in this group will receive the traditional medication only.
  Interventions: Other: Traditional medication

INTERVENTIONS:
Combination Product: Dexamethasone phonophoresis — Ultrasound therapeutic device with the use of 0.4% Dexamethasone sodium phosphate gel for phonophoresis.
  Arms: Group (A)
Device: Laser Acupuncture — low level laser therapy placed in contact with the skin perpendicular over the body acupoints (LI 4) - (LI 20) - (EX- HN5) - (GV 20) - (GV 24) - (ST3) - (ST 7) in both sides and on (EX-HN3) acupoint,
  Arms: Group (B)
Other: Traditional medication — Each participant in this group receive the traditional medication.

SUMMARY:
This study is designed to provide a comprehensive overview of evidence concerning the efficacy and safety of dexamethasone phonophoresis and laser acupuncture for treatment of chronic rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 30 to 50 years.
* Male and female patients will participate in the study.
* All patients have chronic rhinosinusitis, who are experiencing 12 weeks or longer of 2 or more of the following signs and symptoms:

mucopurulent drainage (anterior, posterior, or both) nasal obstruction (congestion) facial pain-pressure-fullness, or decreased sense of smell

• All patients enrolled in the study will have their informed consent.

Exclusion Criteria:

* Patients with metal implants (pacemakers, dental implants, or any other implants).
* Patients with cancer, pregnancy or impaired vascular circulation.
* Patients who suffer from mental or psychological disorders.
* Patients with any systemic diseases that may interfere with the objectives of the study.
* Patients with long-term use of corticosteroids or immunosuppressive agents.
* Congenital defects on face and nose.
* Fracture of nose or face.
* Patients who are contraindicated for corticosteroids use in patient who will receive dexamethasone phonophoresis.
* Allergic patients.
* Pervious nasal surgery.
* Patients with nasal septum deviation.
* patients who had used antihistamines within 1 week, topical corticosteroids within2 weeks, systemic corticosteroids within 4 weeks, anti-cholinergic drugs within 3 days, antileukotriene drugs within 1 week, decongestants within 3 days, tricyclic antidepressants or phenothiazines within 2 weeks, non-steroidal analgesics within 2 weeks or any medication that may interfere with the objectives of the study.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Sino nasal Outcome Test 22 (SNOT-22) | one month
  This is a Quality Of Life Questionnaire specifically designed for sinusitis patient. It consists of 22 item sinus specific question which has to be administered to the patient and the total sum of all the items will be recorded based on the severity of the patient's condition and the scores will be calculated
Computerized Tomography Scan | one month
  CT scan will be used for assessment of mucosal thickening of maxillary sinuses, which is based on 0-3 system: 0 = clear, 1= mild or moderate mucosal thickening, 2 = severe mucosal thickening, 3 = total opacification

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Abd Elaziem Abd Elaziz Walaa Abd Elaziem Abd Elaziz, Doctoral degree, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical therapy, Cairo University, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
pre and post assessment measures results of:
  1. Sino nasal Outcome Test 22 (SNOT-22)
  2. Computerized Tomography Scan:

REFERENCES:
- [Background] da Silva GS, Dos Santos Isoppo K. Therapeutic ultrasound as a treatment for chronic rhinosinusitis: A systematic review. Clin Respir J. 2021 Dec;15(12):1275-1285. doi: 10.1111/crj.13441. Epub 2021 Aug 29. PMID 34423908
- [Background] Lee B, Kwon CY, Park MY. Acupuncture for the Treatment of Chronic Rhinosinusitis: A PRISMA-Compliant Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2022 Aug 31;2022:6429836. doi: 10.1155/2022/6429836. eCollection 2022. PMID 36091598
- [Background] Naghdi S, Ansari NN, Varedi M, Fathali M, Zarrin M, Kashi-Alashti M, HasanNia F. Use of low-level laser therapy for patients with chronic rhinosinusitis: a single-blind, sham-controlled clinical trial. Lasers Med Sci. 2022 Dec 20;38(1):5. doi: 10.1007/s10103-022-03684-z. PMID 36538169